CLINICAL TRIAL: NCT02396225
Title: Concentrations of Voriconazole in Blood and BAL-fluid After Inhalation and Oral Administration
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: results obtained at interrim analysis after 12 patients would not be changed by recruiting another twelwe participants
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: M-2013-242-13
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Invasive Aspergillosis
Keywords: voriconazole; inhalation; aerosol; epithelial lining fluid; concentration; pharmacokinetic
MeSH Terms: conditions — Respiratory Aspiration | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled voriconazole (Experimental): 12 patients inhale voriconazole 40 mg b.i.d for two days
  Interventions: Drug: Voriconazole
- Oral Voriconazole (Active Comparator): 12 patients ingest voriconazole tablets 400 mg b.i.d for one day followed by 200 mg b.i.d for one day
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole

SUMMARY:
Concentrations of voriconazole in pulmonary epithelial lining fluid and in serum are compared after inhalation of 40 mg voriconazole b.i.d. for two days or oral intake of voriconazole tablets 400 mg bid for 1 day followed by 200 mg b.i.d. for one day, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Planned bronchoscopy in relation to work-up after hemoptysis or other symptom leading to bronchoscopy
* Informed written consent
* Performance status 0-1
* Ct scan of thorax without suspicion of malignancy
* Weight t ≥ 60 og ≤ 130 kg
* Male gender or female gender in postmenopausal state defined by amenorrhea in more than 12 months.

Exclusion Criteria:

* Voriconazole treatment up to one week before inclusion
* Se-creatinin≥ 100 uM
* ALAT ≥ 70 U/l
* QT-interval > 480 ms
* Allergic reaction to voriconazole or constituents in Vfend
* Allergic reaction to other azoles
* Ischemic Heart disease, Heart failure or uncontrolled hypertension
* Treatment with statins or omeprazole, which cannot be paused for three days during voriconazole exposure
* Treatment with Efavirenz, rifabutin, ritonavir, everolimus, methadon, alfentanil, fentanyl, sufentanil, oxycodone, hydrocodone, fluconazole, aztemizol, cisaprid, pimozid, quinidine, terfenadine, carbamazepine, phenobarbital, mephobarbital, ergotamine, dihydroergotamine, rifampicine, st. johns worth, everolimus, phenytoin, warfarin, phenprocoumon, acenocoumarol, benzodiazepines as midazolam, triazolam, alprazolam, sirolimus, cyclosporine, tacrolimus, ibuprofen, diclofenac,tolbutamide, glipizide, vincristine, vinblastine or other vinca alkaloids, HIV-protease Inhibitors e.g. saquinavir, amprenavir and nelfinavir, delavirdine, nivrapine and other non-nocleaoside revers transcriptase inhibitors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Voriconazole concentration in serum | 2 years

SECONDARY OUTCOMES:
Voriconazole concentration in lunge epithelial lining fluid | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus C, Denmark